CLINICAL TRIAL: NCT04930679
Title: A Phase I, Open-label Safety Evaluation of Andiabet of Traphaco J.S.C on Diabetes Mellitus Type II
Brief Title: Evaluating Safety of Andiabet on Diabetes Mellitus Type II Patients, Phase I CT.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre of Clinical Pharmacology, Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNLS/2018-03
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 20 diabetes type 2 patients are recruited, in which 14 took part in the study, randomly divided into 2 arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental): 1 capsule of Andiabet x 3 times/ day . Taken 30 minutes before meals in 28 days
  Interventions: Drug: Andiabet
- Group II (Experimental): 2 capsule of Andiabet x 3 times/ day . Taken 30 minutes before meals in 28 days
  Interventions: Drug: Andiabet

INTERVENTIONS:
Drug: Andiabet — Each hard capsule includes: 200mg Gynostemma Pentaphyllum Leaf, 200mg Largerstroemia Speciosa Leaf, 133mg Anemarrhena Asphodeloides Whole

SUMMARY:
This phase I clinical trial is used to evaluate the safety of Andiabet, a herbal-derived medicinal product that assists in the treatment of type 2 Diabetes (T2D). Thereby, determine efficacy of the drug on stabilizing blood glucose in T2D patients.

DETAILED DESCRIPTION:
This is a 28-day phase I, open-label clinical trial to evaluate safety of Andiabet on . The general purpose is the evaluate safety via adverse events and tolerability of Andiabet on T2D patients, and evaluate effect of Andiabet on clinical and laboratory parameters.

The study conducted on volunteering T2D patients, whose HbA1c level is =< 7.5% and are not pregnant, had no records of addiction, allergy, hypersensitivity, and chronic diseases. The main evaluation criteria are fasting glucose, used for evaluating efficacy and safety, which evaluated based on adverse events.

Ensuring quality of the data:

Sponsor and CRO are supervisors. Supervision will be conducted periodically, ensuring the compliance with the research proposal, following GCP.

Hanoi Medical University-Clinical center of Pharmacology is responsible for managing the data. Completed CFR are sent to the Center of Clinical Pharmacology, entered by Microsoft Excel and analysed using SPSS 16.0 Before analysing, these data will be checked randomly, avoiding errors in data entry.

ELIGIBILITY:
Inclusion Criteria: Participants must meet ALL the following criteria:

* Type 2 Diabetes (T2D) patients with HbA1c lower than or equal to 7.5%
* BMI range: 18-40 kg/m2
* Diagnosed with T2D or currently treating T2D (prescribed by physicians) with one or more of the following drugs: Metformin, Sulfonyl urea, dipeptidyl peptidase-4 inhibitors, or a-glucosidase inhibitors
* Be able to stop using T2D drugs in 4 weeks, while maintaining diets and exercising routine.
* Willing to take part in the study.

Exclusion Criteria: Participants that have ONE of the following:

* Diagnosed with Type 1 Diabetes.
* History of complications due to Diabetes Mellitus.
* History of cardiovascular diseases: hypertension, heart failure, Unstable agina, stroke or transient ischemic attack, myocardial infarction, arrhythmias, coronary artery interventions.
* History of drugs, alcohol addiction.
* Uncontrolled high blood pressure
* Pre-study screening blood test with abnormal results in total blood compositions, urea, AST, ALT, creatinine, albumin, total bilirubin, total urine analysis.
* Test positive for HIV or HbsAg
* Abnormal ECG results that are clinically significant.
* History of hypersensitivity to any of the ingredients in the testing product.
* Female participants that are pregnant or having pregnancy intention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-24 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Adverse events | 28 days
  2 AEs recorded, there were changes in biochemical indices. However, these AEs are considered mild and unrelated to the investigated product.
Fasting blood glucose | 28 days
  Group II is reported to have lower blood glucose compared to group I. However, the difference is efficacy is not clear between 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Dung C Nguyen, MD, Principal Investigator — Center of Clinical Pharmacology, Hanoi Medical University
Locations (1):
- Centre of Clinical Pharmacology, Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No